CLINICAL TRIAL: NCT00923533
Title: An Open-label, Multiple-dosing, Crossover, and Parallel Study to Evaluate the Safety and Pharmacokinetics After Oral Concurrent Administration of Fimasartan and Hydrochlorothiazide in Healthy Male Volunteers
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics After Oral Concurrent Administration of Fimasartan and Hydrochlorothiazide in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Choi, Director, Boryung Pharm Co., Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: A657-BR-CT-103
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Essential Hypertension
Keywords: Fimasartan; Drug interaction
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Active Comparator): Fimasartan (7day) Fimasartan + Hydrochlorothiazide (7day)
  Interventions: Drug: Fimasartan
- Part B (Active Comparator): Hydrochlorothiazide (7day) Hydrochlorothiazide + Fimasartan (7day)
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Fimasartan — Fimasartan (7day) Fimasartan + Hydrochlorothiazide (7day)
  Arms: Part A
Drug: Hydrochlorothiazide — Hydrochlorothiazide (7day) Fimasartan + Hydrochlorothiazide (7day)
  Arms: Part B

SUMMARY:
To evaluate drug-drug interaction between fimasartan and hydrochlorothiazide.

DETAILED DESCRIPTION:
Fimasartan (BR-A-657-K), a selective blocker of AT1 receptor subtype, showed the rapid and potent antihypertensive effect in many hypertensive models.

Phase I study, Fimasartan (BR-A-657-K) 20 mg ~ 480 mg single dosing with healthy subjects, demonstrated that the Fimasartan (BR-A-657-K) was very safe and well tolerated. Another phase I study, Fimasartan (BR-A-657-K) 120mg and 360mg dosing for 7 days, also showed that Fimasartan (BR-A-657-K) was safe and tolerable though one temporal adverse event was observed in high dose.

A open-labeled, multiple-dosing, crossover, parallel Clinical Study to Evaluate drug-drug interaction between fimasartan and hydrochlorothiazide.

34 male healthy volunteers were enrolled during 2 months.

In part A, 240 mg of fimasartan per day was taken for 1 week. After 7 day washout period, 240 mg of fimasartan and 25mg of hydrochlorothiazide per day were taken for 1 week. Then blood and urine samples were collected 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours at 7 day and 21 day.

In part B, 25 mg of hydrochlorothiazide per day was taken for 1 week. After 7 day washout period, 240 mg of fimasartan and 25mg of hydrochlorothiazide per day were taken for 1 week. Then blood and urine samples were collected 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours at 7 day and 21 day.

ELIGIBILITY:
Inclusion Criteria:

* age: 20 - 45 years
* sex: male
* body weight: greater than 55 kg
* written informed consent

Exclusion Criteria:

* known allergy to Fimasartan and hydrochlorothiazide
* existing cardiac or hematological diseases
* existing hepatic and renal diseases
* existing gastrointestinal diseases
* acute or chronic diseases which could affect drug absorption or metabolism
* history of any serious psychological disorder
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day 3 month ago
* participation in a clinical trial during the last 2 months prior to the start of the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
AUC, Cmax, Tmax, CL/F | 0, 0.5, 1, 1.5, 2, 2.5 3, 4, 6, 8, 12, 24 hours at 7 day and 21 day

REFERENCES:
- [Derived] Gu N, Kim BH, Lim KS, Kim SE, Nam WS, Yoon SH, Cho JY, Shin SG, Jang IJ, Yu KS. The effect of fimasartan, an angiotensin receptor type 1 blocker, on the pharmacokinetics and pharmacodynamics of warfarin in healthy Korean male volunteers: a one-sequence, two-period crossover clinical trial. Clin Ther. 2012 Jul;34(7):1592-600. doi: 10.1016/j.clinthera.2012.06.004. Epub 2012 Jun 22. PMID 22727611